CLINICAL TRIAL: NCT04895540
Title: South Asian Arrhythmogenic Cardiomyopathy Registry
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sheri Kashmir Institute of Medical Sciences (Other)
Collaborators: Indian Heart Rhythm Society (Unknown); Sri Jayadeva Institute of Cardiovascular Sciences and Research (Other); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Dr Muzaffar Ali, Principal Investigator, Sheri Kashmir Institute of Medical Sciences
Other Study IDs: SKIMSCL-2021-001
Record Dates: First submitted 2021-05-17; First posted 2021-05-20 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Arrhythmogenic Right Ventricular Cardiomyopathy; Arrhythmogenic Right Ventricular Dysplasia; Arrhythmogenic Ventricular Cardiomyopathy; Arrhythmogenic Cardiomyopathy; Ventricular Tachycardia; Sudden Cardiac Death
MeSH Terms: conditions — Arrhythmogenic Right Ventricular Dysplasia; Tachycardia, Ventricular; Death, Sudden, Cardiac | interventions — Electrocardiography; Echocardiography; Genetic Testing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — Blood samples Buccal swab
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Diagnosed ACM patients
  Interventions: Diagnostic Test: ECG; Diagnostic Test: Echocardiography; Diagnostic Test: Cardiac MRI; Diagnostic Test: Ambulatory ECG recording; Diagnostic Test: Cardiac EP study; Genetic: All study subjects will undergo sample collection for genetic testing.
- First degree relatives of ACM patients
  Interventions: Diagnostic Test: ECG; Diagnostic Test: Echocardiography; Genetic: All study subjects will undergo sample collection for genetic testing.
- Relatives of ACM patients who have suffered an SCD
  Interventions: Diagnostic Test: ECG; Diagnostic Test: Echocardiography; Genetic: All study subjects will undergo sample collection for genetic testing.

INTERVENTIONS:
Diagnostic Test: ECG — All study subjects will undergo ECG recording.
Diagnostic Test: Echocardiography — All study subjects will undergo transthoracic echocardiography
Diagnostic Test: Cardiac MRI — All ACM patients and SCD survivors will undergo cardiac MRI testing.
  Groups: Diagnosed ACM patients
Diagnostic Test: Ambulatory ECG recording — All ACM patients and SCD survivors will undergo 24-hour ambulatory ECG recording
  Groups: Diagnosed ACM patients
Diagnostic Test: Cardiac EP study — ACM patients and SCD survivors will undergo diagnostic cardiac Electrophysiology testing.
  Groups: Diagnosed ACM patients
Genetic: All study subjects will undergo sample collection for genetic testing. — Blood samples and buccal swab will be collected from study subjects for genetic testing.

SUMMARY:
Arrhythmogenic Cardiomyopathy (ACM) is increasingly identified as an important cause of cardiac morbidity and mortality, especially of SCD, in a younger population.

Although there are no epidemiological data available, the investigators' experience is that in the North Indian region, ACM is rare outside our regions. ACM is also an understudied cardiac disorder in the South-Asian region.

An ethnic nonmigratory population inhabits the two regions, and consanguineous marriages are common. Based on these observations, the investigators firmly believe that there may be a founder gene in our populations responsible for the increased incidence of ACM.

Our project includes a thorough phenotypic analysis ((ECG, Holter, and echocardiography) in the ACM patients and their first-degree relatives; cardiac MRI and high resolution endocardial bipolar and unipolar voltage mapping (using HD grid catheter) in the patients.

The patient provided blood for the extraction of DNA will first undergo target panel sequencing for 20 known classic right-dominant ACM and left-dominant ACM. If this is negative for known pathogenic and likely pathogenic variants but identified novel variants of uncertain significance (VUS), then co-segregation analysis in family members will be performed. This technique can provide helpful information to reclassify VUSs. If both these are negative, then whole-exome 'trio' analysis will be performed, whch includes the proband and two family members, to triangulate from all 20,000 genes to a list of candidates for further interrogation.

The investigators wish to provide comprehensive answers to the research question by combining the genetic analysis with phenotypic evaluation.

DETAILED DESCRIPTION:
Arrhythmogenic Cardiomyopathy (ACM) is an inherited cardiomyopathy characterized by structural and functional abnormalities in the right ventricle (and left ventricle, in 50%) resulting in ventricular arrhythmias.1 It is an important cause of sudden cardiac death (SCD) in young adults, accounting for 11% of all cases.2 The hallmark lesion of ACM is replacement of the ventricular myocardium by fibrofatty tissue. 3ARVC is most often familial, with autosomal dominant inheritance, autosomal recessive inheritance being uncommon. However, in relatively isolated populations, autosomal recessive forms are recognized and often have more severe phenotype. In fact, the first two genes discovered for ARVC were Naxos and Carvajal syndromes, in isolated populations of Naxos Island and Equadorian populations respectively.

The genes involved in the pathogenesis of ACM are most often desmosomal genes like plakoglobin (JUP), desmoplakin (DSP), plakophilin-2 (PKP2), desmoglein-2 (DSG2), desmocollin-2 (DSC2). PKP2 mutations are the most common. However, there are disease-causing genes that cause "classic" right ventricular ACM that do not encode for desmosomal proteins.4 The term "ALVC" has been proposed to recognize ACM of LV origin as distinct from right ventricular ACM in which there is predominantly LV arrhythmia and structural abnormalities.4 The most common clinical presentation consists of ventricular arrhythmias and related symptoms/events, which include palpitations, syncopal episodes (mostly occurring during physical exercise), and cardiac arrest. The diagnosis of biventricular or predominant left AC may be missed at the onset of symptoms in some patients who present years later with heart failure, with or without ventricular arrhythmias, and are incorrectly diagnosed as having idiopathic dilated cardiomyopathy.5 The diagnosis of ACM is based on the 2010 Task Force Criteria (TFC), which include repolarization abnormalities, depolarization abnormalities, arrhythmias, tissue characterization, structural abnormalities, and family history. However, there is no agreed gold-standard, and limitations of the Task Force Criteria are: a) the sentinel event can be SCD, with very subtle morphological abnormalities, which may not be identified at post-mortem examination b) Electrical abnormalities can precede the structural abnormalities, which can be easily missed. This has a huge impact on family members, as they do not undergo appropriate clinical or genetic testing - missing an opportunity to intervene and save lives c) Disease expression in the pediatric population is uncommon d) the long list of criteria and modalities in the TFC make diagnosing ACM complex and time-consuming. Identifying novel gene mutations in ACM may help in further understanding the pathogenesis of the disease and may help in finding a new pharmacological target for such patients.

i. Design of the study Prospective, cohort study

ii. Inclusion and exclusion criteria

Inclusion criteria:

Patients diagnosed with ACM according to 2010 Task Force Criteria Parents of ACM patients Siblings of ACM patients Relatives of ACM patients who have suffered an SCD

Exclusion criteria:

ACM patients or their relatives refuse to give consent for participation in the study. Study subjects who refuse to provide consent for a specific test or investigation will not be excluded.

iii. Endpoints:

1. Patients: Completion of the following data collection of all the patients:

   ECG, Holter, Echocardiography, cardiac MRI, Endocardial voltage mapping, genetic analysis along with blood and buccal samples for genetic analysis
2. Parents/siblings: Completion of the following data of all the parents, siblings: ECG, Echocardiography along with blood and buccal samples for genetic analysis
3. SCD affected relatives of ACM patients: Completion of the following data of the affected relatives: ECG, Holter, Echocardiography, cardiac MRI along with blood and buccal samples for genetic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with ACM according to 2010 Task Force CriteriaParents of ACM patients
* Siblings of ACM patients
* Relatives of ACM patients who have suffered an SCD

Exclusion Criteria:

* ACM patients or their relatives who refuse to give consent for participation in the study.
* Study subjects who refuse to provide consent for a specific test or investigation will not be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population will consist of ACM patients and their first degree relatives and other relatives who have suffered an SCD
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-04-10 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Completion of Data collection and phenotypic evaluation | May 2021-April 2022
Completion of genetic analysis | May 2021-April 2022
Phenotypic and genotpic assessment | May 2022-June 2022

CONTACTS AND LOCATIONS:
Locations (3):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States
- India (2):
  - Sher-i-Kashmir Institute of Medical Sciences, Srinagar, Jammu and Kashmir
  - Sri Jayadeva Institute of Cardiovascular Sciences and Research, Bangalore, Karnataka

IPD SHARING:
Plan to Share IPD: No